CLINICAL TRIAL: NCT02625870
Title: A 12-Week, Randomized, Double-Blind, Corn Oil-Controlled Phase 3 Study to Assess the Efficacy and Safety of Omega-3-Acid Ethyl Esters 90 Soft Capsules in Subjects With Severe Hypertriglyceridemia
Brief Title: Omega-3-Acid Ethyl Esters 90 Soft Capsules for Lowering Very High Triglycerides
Acronym: OMEELVHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HROMEE2015
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3-Acid Ethyl Esters 90 Soft Capsules (Experimental)
  Interventions: Drug: Omega-3-Acid Ethyl Esters 90 Soft Capsules
- Corn Oil (Placebo Comparator)
  Interventions: Drug: Corn Oil

INTERVENTIONS:
Drug: Omega-3-Acid Ethyl Esters 90 Soft Capsules — Omega-3-Acid Ethyl Esters 90 Soft Capsules will be provided in 1 g polyacrylate-coated soft gel capsules.Four capsules will be taken with breakfast once per day, for 12 weeks.
  Arms: Omega-3-Acid Ethyl Esters 90 Soft Capsules
Drug: Corn Oil — Corn Oil will be provided in 1 g polyacrylate-coated soft gel capsules.Four capsules will be taken with breakfast once per day, for 12 weeks.
  Arms: Corn Oil

SUMMARY:
The trial was a double-blind, randomized, parallel-group study comparing Omega-3-Acid Ethyl Esters 90 Soft Capsules and placebo. The primary objective of the present study was to evaluate the efficacy and safety of Omega-3-Acid Ethyl Esters 90 Soft Capsules in subjects with severe hypertriglyceridemia (TGs ≥500 mg/dL but <2000 mg/dL).

ELIGIBILITY:
Inclusion Criteria:

-1.At least 2 times of fasting serum TG concentrations≥500 mg/dL but<2000 mg/dL at screening (2and 1 and 0 weeks before random assignment).

2.Two times qualified High Triglycerides Dietary Assessment Table at 2 and 0 weeks before random assignment according to the "prevention and treatment of dyslipidemia in Chinese adults Guide ".

Exclusion Criteria:

* 1.Unable to discontinue use of other omega-3 fatty acid-containing products, bile acid sequestrants, fibrates ,niacin or any supplement used to alter lipid metabolism throughout the entire study.

  2.Patients taking bile acid sequestrants, fibrate, niacin or any supplement used to alter lipid metabolism more than 6 weeks before entering the study dietary phase.

  3.Subjects consuming omega-3 fatty acid-containing products such as cod liver oil, or lipid-decreasing fibers at least 4 weeks before beginning the study.

  4.Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>3 times the upper limit of normal.

  5.Serum creatinine >176μmol/L. 6.Platelet counts<60×109/L，hemoglobin <100 g/L. 7.Poorly controlled hypertension(resting blood pressure ≥160 mm Hg systolic or ≥100 mm Hg diastolic) 8.Uncontrolled type II diabetes(fasting blood sugar >11.1mmol/L). 9.Type II diabetes, nephrotic syndrome, hypothyroidism. 10.Atrial fibrillation. 11.History of pancreatitis and symptomatic gallstone disease, unless treated with cholecystectomy.

  12.History of cancer (other than basal cell carcinoma) in the past 2 years. 13.Allergy or intolerance to omega-3 fatty acids, omega-3-acid ethyl esters, or fish.

  14.History in the past 12 months of drug abuse or alcohol abuse (.14 drinks per week; 1 drink was equivalent to 12 oz beer, 5 oz wine, or 1.5 oz hard liquor) was also exclusionary.

  15.Exposure to any investigational product, within 30 days prior to Visit. 16.Presence of any other condition the Investigator believes would interfere the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
End-of-treatment Serum Triglycerides percentage change from baseline under fasting conditions | 12 weeks

SECONDARY OUTCOMES:
End-of-treatment non-HDL-C percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment TC percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment VLDL-C percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment HDL-C percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment LDL-C percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment LDL-C/HDL-C percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment Apo A5 percentage change from baseline under fasting conditions | 12 weeks
End-of-treatment Apo C3 percentage change from baseline under fasting conditions | 12 weeks